CLINICAL TRIAL: NCT05988632
Title: Intranasal Insulin for Treatment of Alcohol Use Disorder
Acronym: ITA
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Responsible Party: Principal Investigator, Carolina L Haass-Koffler, Associate Professor, Brown University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00000134
Record Dates: First submitted 2023-07-25; First posted 2023-08-14 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Insulin, Then Placebo (Experimental): There will be one single administration of intranasal human insulin (80IU) before alcohol self-administration. After a one week washout period, there will be one single intranasal administration of placebo (saline, 0.9% solution) before alcohol self administration.
  Interventions: Drug: Regular Human Insulin then Placebo
- Placebo, Then Insulin (Experimental): There will be one single intranasal administration of placebo (saline, 0.9% solution) before alcohol self administration. After a one week washout period, there will be one single administration of intranasal human insulin (80IU) before alcohol self-administration.
  Interventions: Drug: Placebo then Regular Human Insulin

INTERVENTIONS:
Drug: Regular Human Insulin then Placebo — Insulin: 80 IU (administered intranasally) THEN Placebo: 0.9% saline solution (administered intranasally)
  Other Names: Novolin R
  Arms: Insulin, Then Placebo
Drug: Placebo then Regular Human Insulin — Placebo: 0.9% saline solution (administered intranasally) THEN Insulin: 80 IU (administered intranasally)
  Other Names: Novolin R
  Arms: Placebo, Then Insulin

SUMMARY:
This is a randomized controlled trial (RCT), within-subject, crossover, double-blind, placebo-controlled in non-treatment-seeking individuals with Alcohol Use Disorder (AUD) (N=40, 50% female) randomized to IN insulin or placebo. In a bar laboratory setting, randomized participants will receive a single dose of IN insulin (80IU) or an IN matched placebo (0.9% Saline). Participants will undergo a cue-reactivity paradigm followed by an alcohol challenge that includes an alcohol drink designed to raise the breath alcohol content (BrAC) to 0.08g/dL.

DETAILED DESCRIPTION:
Aims in this RCT testing the effect of IN insulin, compared to placebo, in individuals with AUD include the following:

AIM 1: to assess the safety, tolerability and acceptability of IN insulin as a pharmacological intervention for AUD. The data collected in this aim will monitor possible adverse events and yield qualitative and quantitative data to finalize the feasibility and acceptability of IN insulin as an AUD pharmacotherapy.

Aim 2 (alcohol-drug interaction): to assess the safety and tolerability of IN insulin when administered with alcohol. The investigators will use a battery of physiological/psychological assessments that measures potential adverse events, alcohol subjective response and alcohol pharmacokinetics endpoints.

ELIGIBILITY:
Inclusion Criteria:

* ≥21 years

  * meet any DSM-5 criteria score for AUD
  * Individuals who, in the last month, have consumed at least the same amount of alcohol that will be administered in the laboratory procedure (i.e. to reach BrAC levels of 0.08g/dl, ~two drinks in one occasion)
  * BrAC=0.00g/dL at each visit
  * good health as confirmed by medical history, physical examination and lab tests
  * willing to adhere to the study procedures
  * understand informed consent and questionnaires in English at an 8th grade level
  * willing to have glucose monitored by finger stick during the laboratory procedures

Exclusion Criteria:

* • female identifying who are breastfeeding or pregnant (assessed by a urine screen)

  * individuals with diabetes
  * history of suicide attempts in the last three years
  * current diagnosis of other substance use disorder (other than nicotine or cannabis)
  * use of drugs (e.g. stimulants/opioids) at each alcohol administration session (by urine tox screen)
  * cannabis intoxication (by clinical assessments)
  * use of medications that may interact with insulin and alcohol (by Micromedex database)
  * hypersensitivity to insulin
  * any nasal disease/congestion that may interfere with intranasal drug absorption;
  * baseline hypoglycemia (blood glucose ≤65mg/dL) or hyperglycemia (blood glucose >200mg/dL) (by finger stick)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
intranasal adverse events | From baseline to post-treatment (1 day)
  Adverse event reported during the drug administration

SECONDARY OUTCOMES:
insulin alcohol interaction | From baseline to post-treatment (1 day)
  Adverse event reported during the alcohol administration

CONTACTS AND LOCATIONS:
Locations (1):
- Brown University, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haass-Koffler CL, Kashyap B, Gully BJ, Nambiar SS, Hornbacher R, Foster SL, Silberman Y, Swift RM, Hanson LR, Frey WH 2nd. Intranasal insulin for the treatment of alcohol use disorder: design and methodology of an alcohol interaction randomized controlled trial. Contemp Clin Trials Commun. 2025 Jun 10;46:101509. doi: 10.1016/j.conctc.2025.101509. eCollection 2025 Aug. PMID 40584152